CLINICAL TRIAL: NCT01953497
Title: A Phase I, Placebo-controlled, Randomized, Double Blind, Single or Multiple Dose Study of URC102 in Healthy Male Volunteers of Korean and Caucasian to Assess Safety, Pharmacokinetics and Pharmacodynamics
Brief Title: Phase 1 Study of URC102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: URC001KR
Record Dates: First submitted 2013-09-13; First posted 2013-10-01 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — URC102

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- URC102 (Active Comparator): URC102
  Interventions: Drug: URC102

INTERVENTIONS:
Drug: URC102
  Arms: URC102
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the safety, tolerability, PK and PD of URC102 in healthy subjects. To evaluate the food effect on PK.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Received other investigational drug within 12 weeks prior to the first dose of study drug

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2013-12-24 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with AE | 1 week

SECONDARY OUTCOMES:
Plasma URC102 concentration | 1 week
Blood uric acid | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, MBA, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee HA, Yu KS, Park SI, Yoon S, Onohara M, Ahn Y, Lee H. URC102, a potent and selective inhibitor of hURAT1, reduced serum uric acid in healthy volunteers. Rheumatology (Oxford). 2019 Nov 1;58(11):1976-1984. doi: 10.1093/rheumatology/kez140. PMID 31056705